CLINICAL TRIAL: NCT00957437
Title: A Phase I, Randomised, Open, Single-centre Study to Evaluate the Pharmacokinetics of Different Extended-release Formulations of AZD1305 When Given as Single and Repeated Oral Doses to Healthy Male Volunteers
Brief Title: Study to Assess Drug Concentrations in Plasma of Different Extended-release Formulations of AZD1305
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3190C00016
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Phase 1; healthy volunteer; male; pharmacokinetics; AZD1305
MeSH Terms: interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: 3 way crossover (Experimental): AZD1305: ER test formulation 1 (w/wo food) and reference formulation
  Interventions: Drug: AZD1305
- Part B1: single arm (Experimental): AZD1305: ER test formulation 1
  Interventions: Drug: AZD1305
- Part B2: 3 way crossover (Experimental): AZD1305: ER test formulation 2 (w/wo food) and reference formulation
  Interventions: Drug: AZD1305

INTERVENTIONS:
Drug: AZD1305 — Single Oral Dose, ER formulation 1
  Arms: Part A: 3 way crossover
Drug: AZD1305 — ER formulation 1, bid for 5 days
  Arms: Part B1: single arm
Drug: AZD1305 — Single Oral Dose, ER formulation 2
  Arms: Part B2: 3 way crossover

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of different extended-release formulations of AZD1305 when given as single and multiple oral doses to healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures.
* Body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg.

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder in the opinion of the investigator.
* Use of nicotine in the last 4 weeks before screening and not more than 7 cigarettes per week (equivalent to 1 nicotine patch or 7 nicotine gums per week) before then. There will be no smoking until follow-up visit.
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs or ECG at baseline in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-08; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables of AZD1305 by assessment of drug concentrations in plasma | From predose until 48 hours post last dose

SECONDARY OUTCOMES:
Adverse Events, ECG variables, vital signs, physical examination, laboratory variables and weight | Frequent safety measurements during the study, from screening period to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lunde, Study Director — AstraZeneca R&D, Mölndal, Sweden; Klaus Francke, Principal Investigator — PAREXEL Early Phase Clinical Unit, London UK.
Locations (1):
- Research Site, Harrow, United Kingdom